CLINICAL TRIAL: NCT05535881
Title: Strengths to Grow: An Online Parenting Resource
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Margaret Lumley, Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-08-001
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-07

CONDITIONS: Happiness; Self Efficacy; Positive Affect

STUDY DESIGN:
Intervention Model Description: The current study is a two-wave randomized controlled trial that employs a 2 (group - between participants) by 2 (time - within participants) mixed measures design to assess a brief online strength-based parenting program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Behavioral: Strengths to Grow Program
- Waitlist Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Strengths to Grow Program — In an online, self-directed format, the Strengths to Grow program will present the principles of strength-based parenting using videos, pictures, reflection questions, and written text. The intervention will communicate that a) every child has a unique set of strengths and that b) noticing and developing these strengths can enhance child and family well-being. It will also provide concrete steps that parents can follow to talk with their child about strengths, and it will provide ideas for family activities that would allow family members to express strengths. Participants will be invited to respond to reflection questions at various points throughout the program.
  Arms: Experimental Group

SUMMARY:
Research suggests that strength-based parenting programs can enhance family well-being, but the current formats of these programs (e.g., in-person workshops) are not accessible to many families. The first aim of the study is to develop a strength-based parenting program that is delivered in an accessible and engaging format. A community sample of parents will interact with the online program and complete a brief interview to provide suggestions to increase accessibility and engagement. The second aim of the study is to assess the effectiveness of a strength-based parenting program delivered in an online, interactive format. Toward this end, parents of children in kindergarten to Grade 3 will be invited to complete a brief, online survey of well-being before and a few weeks after completing the online program to assess its impact on well-being.

DETAILED DESCRIPTION:
Strength-based Parenting

Strength-based parenting is a style of caregiving which identifies and cultivates strengths in the child and caregiver. When parents employ a strength-based parenting style, youth tend to demonstrate greater academic achievement, resilience, and overall well-being, and parents tend to experience more well-being within the caregiving role. Additionally, it is believed that caregivers can develop a strength-based parenting style through training and practice. For these reasons, several strength-based parenting programs have been developed.

Character Strengths

Strength-based parenting programs typically focus on helping parents to identify and develop a particular type of strength known as character strengths. Character strengths are personal qualities that are widely regarded as morally good (e.g., bravery, curiosity, kindness). In 2004, Peterson and Seligman completed a comprehensive review that identified 24 character strengths. The development and use of these 24 character strengths has consistently been shown to be associated with well-being across the lifespan.

Strength-based Parenting Programs

The content of strength-based parenting programs typically revolves around introducing parents to character strengths, helping parents to identify character strengths within themselves and their child, teaching parents to notice and encourage their child's use of strengths, and helping parents to employ their strengths within the caregiving role. Within the published literature, strength-based parenting programs have been delivered in two formats: in-person workshops and online handouts. These programs had positive effects, including improving caregiving self-efficacy, positive emotions toward the child, and family well-being relative to waitlist control groups. However, the format of these programs may have limited the number of parents who could access and engage with the resources.

Access and Engagement

It is important to consider the extent to which caregivers can access and engage with programs because access and engagement are necessary pre-requisites to program effectiveness. Research on parenting programs suggests that in-person workshops are not accessible to many families, particularly families of lower socio-economic status. Online handouts may be more accessible, but may struggle to engage families, as interactive, media-rich online materials tend to be more engaging. The present study aims to increase the accessibility of strength-based parenting programs by offering the resources online, and to increase engagement by providing interactive rather than static online materials.

An Online, Interactive, Strength-based Parenting Program

O'Byrne et al. examined pilot project data from an online, interactive strength-based parenting program. The thirty-minute program was delivered to parents of kindergarten children. Through focus groups and analyzing parents' interactions with the online program, the pilot project found that parents reacted positively to the online, interactive format and the strength-based content. Additionally, within the sample, the program was accessible to families of lower socio-economic status who are difficult to access with in-person resources. Although the pilot project generated promising results, it relied on a small sample and effectiveness was not examined. The present project aims to build upon this initial work by using the pilot project results to revise the program and evaluating the revised program using a larger sample of caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child(ren) who is enrolled in Kindergarten to Grade 3 at the Upper Grand District School Board in Guelph, Ontario
* Able to read and write in English (linguistic proficiency equivalent to a Grade 8 reading level or greater)
* Consent to participate in the research study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Parenting Sense of Competence Scale: Efficacy Subscale | 1 week
  The efficacy subscale of the Parenting Sense of Competence Scale (PSOC) is a 7-item measure of caregivers' perceived competence and capability in handling child problems (e.g., "I honestly believe I have all the skills necessary to be a good parent to my child"). Participants respond to each item using a 6-point scale ranging from strongly disagree to strongly agree. Total scores range from 7 to 42 with higher scores indicate higher caregiving self-efficacy.
Modified Differential Emotions Scale | 1 week
  The Modified Differential Emotions Scale (mDES) is a ten-item measure of the frequency of positive emotions. Participants rate how often they have felt a particular positive emotion (e.g., grateful) in the past two weeks using a 5-point scale ranging from "never" to "most of the time". Consistent with Waters and Sun (2016), the scale instructions will be modified to assess the frequency of positive emotions felt in relation to the parents' child (i.e., "Thinking about your child(ren), how often do you feel each of the following?") Total scores range from 10 to 50 with higher scores indicate more positive emotions toward the child(ren).
Subjective Happiness Scale | 1 week
  The four-item Subjective Happiness Scale (SHS) assesses participant's sense of their overall well-being. Participants respond to items (e.g., Some people are generally very happy. They enjoy life regardless of what is going on, getting the most out of everything. To what extent does this characterization describe you?) on a 7-point scale that differs across items. Total scores range from 4 to 28 with higher scores indicate higher happiness.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lumley, PhD, CPsych, Principal Investigator — University of Guelph
Locations (1):
- Upper Grand District School Board, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data as this has not been approved by our Research Ethics Board.

REFERENCES:
- [Background] Danaher BG, Boles SM, Akers L, Gordon JS, Severson HH. Defining participant exposure measures in Web-based health behavior change programs. J Med Internet Res. 2006 Aug 30;8(3):e15. doi: 10.2196/jmir.8.3.e15. PMID 16954125
- [Background] Eisner M, Meidert U. Stages of parental engagement in a universal parent training program. J Prim Prev. 2011 Apr;32(2):83-93. doi: 10.1007/s10935-011-0238-8. PMID 21424399
- [Background] Fernandez MA, Eyberg SM. Predicting treatment and follow-up attrition in parent-child interaction therapy. J Abnorm Child Psychol. 2009 Apr;37(3):431-41. doi: 10.1007/s10802-008-9281-1. PMID 19096926
- [Background] Fredrickson, B. L. (2013). Chapter One-Positive Emotions Broaden and Build. In P. Devine & A. Plant (Eds.), Advances in Experimental Social Psychology (Vol. 47, pp. 1-53). Academic Press. https://doi.org/10.1016/B978-0-12-407236-7.00001-2
- [Background] Ivtzan, I., Niemiec, R. M., & Briscoe, C. (2016). A study investigating the effects of Mindfulness-Based Strengths Practice (MBSP) on wellbeing. International Journal of Wellbeing, 6(2), 1-13. https://doi.org/10/gfscgj
- [Background] Jach, H. K., Sun, J., Loton, D., Chin, T.-C., & Waters, L. (2018). Strengths and subjective wellbeing in adolescence: Strength-based parenting and the moderating effect of mindset. Journal of Happiness Studies, 19(2), 567-586. https://doi.org/10/gfscg9
- [Background] Johnston, C., & Mash, E. J. (1989). A Measure of Parenting Satisfaction and Efficacy. Journal of Clinical Child Psychology, 18(2), 167-175. https://doi.org/10.1207/s15374424jccp1802_8
- [Background] Kazdin, A. E., & Rabbitt, S. M. (2013). Novel models for delivering mental health services and reducing the burdens of mental illness. Clinical Psychological Science, 1(2), 170-191. https://doi.org/10/gc4pnm
- [Background] Lavigne JV, Lebailly SA, Gouze KR, Binns HJ, Keller J, Pate L. Predictors and correlates of completing behavioral parent training for the treatment of oppositional defiant disorder in pediatric primary care. Behav Ther. 2010 Jun;41(2):198-211. doi: 10.1016/j.beth.2009.02.006. Epub 2009 Dec 5. PMID 20412885
- [Background] Lyubomirsky, S., & Lepper, H. S. (1999). A Measure of Subjective Happiness: Preliminary Reliability and Construct Validation. Social Indicators Research, 46(2), 137-155. https://doi.org/10.1023/A:1006824100041
- [Background] McGoron, L., & Ondersma, S. J. (2015). Reviewing the need for technological and other expansions of evidence-based parent training for young children. Children and Youth Services Review, 59, 71-83. https://doi.org/10/f8bhbv
- [Background] O'Byrne R, Thompson R, Friedmann JS, Lumley MN. Parent Engagement with an Online, School-Based, Character Strengths Promotion Program. Int J Appl Posit Psychol. 2022;7(3):355-377. doi: 10.1007/s41042-022-00072-4. Epub 2022 Aug 11. PMID 35971433
- [Background] Peterson, C., & Seligman, M. E. P. (2004). Introduction to a "manual of the sanities." In Character strengths and virtues (pp. 18-104). American Psychological Association; Oxford University Press. https://books.scholarsportal.info/uri/ebooks/ebooks0/oxford/2009-11-30/3/0195167015
- [Background] Ritterband, L. M., Cox, D. J., Gordon, T. L., Borowitz, S. M., Kovatchev, B. P., Walker, L. S., & Sutphen, J. L. (2006). Examining the Added Value of Audio, Graphics, and Interactivity in an Internet Intervention for Pediatric Encopresis. Children's Health Care, 35(1), 47-59. https://doi.org/10.1207/s15326888chc3501_5
- [Background] Shoshani A, Shwartz L. From Character Strengths to Children's Well-Being: Development and Validation of the Character Strengths Inventory for Elementary School Children. Front Psychol. 2018 Nov 2;9:2123. doi: 10.3389/fpsyg.2018.02123. eCollection 2018. PMID 30450070
- [Background] Waters, L. (2015a). The relationship between strength-based parenting with children's stress levels and strength-based coping approaches. Psychology, 06(06), 689-699. https://doi.org/10/gdj4w6
- [Background] Waters, L. (2015b). Strength-based parenting and life satisfaction in teenagers. Advances in Social Sciences Research Journal, 2(11), 158-173. https://doi.org/10.14738/assrj.211.1651
- [Background] Waters, L. (2020). Using positive psychology interventions to strengthen family happiness: A family systems approach. The Journal of Positive Psychology, 0(0), 1-8. https://doi.org/10.1080/17439760.2020.1789704
- [Background] Waters, L., Loton, D., & Jach, H. K. (2018). Does Strength-Based Parenting Predict Academic Achievement? The Mediating Effects of Perseverance and Engagement. Journal of Happiness Studies. https://doi.org/10/gfscg8
- [Background] Waters, L., & Sun, J. (2016). Can a brief strength-based parenting intervention boost self-efficacy and positive emotions in parents? International Journal of Applied Positive Psychology, 1(1), 41-56. https://doi.org/10/gfschb